CLINICAL TRIAL: NCT01447069
Title: Use of Beta-agonists in Stable Severe Congestive Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTA-HF-01
Record Dates: First submitted 2011-09-25; First posted 2011-10-05 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-08

CONDITIONS: Ischemic Cardiomyopathy; Non-ischemic Cardiomyopathy; Heart Failure
Keywords: heart failure stage 3; beta 2 agonist; N-terminal pro-brain natriuretic peptide; ejection fraction <35%
MeSH Terms: conditions — Heart Failure | interventions — Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Salbutamol (Active Comparator): The patients in the study groups will receive the selective β2 agonist, Salbutamol, in addition to their ongoing optimal heart failure therapy.
  Interventions: Drug: Salbutamol
- control (No Intervention): The patients in the control group will continue with their regular optimal medical therapy without any intervention.

INTERVENTIONS:
Drug: Salbutamol — The initial dose will be 0.5mg bid, with acceleration of the dose every two weeks by 1mg, up to a maximal dose of 2mg bid or an increase in heart rate by 50% above the baseline heart rate, as long as it remains <100 bpm
  Arms: Salbutamol

SUMMARY:
The purpose of this study is to determine whether Salbutamol is effective in the treatment of severe heart failure due to ischemic and non- ischemic cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory Patients with a diagnosis of ischemic and non-ischemic cardiomyopathy with a measured EF <35%, class III as defined by the NYHA with ICD and who receive optimal pharmacological therapy.

Exclusion Criteria:

* Heart Failure class I, II, IV
* atrial fibrillation
* any significant valvular disease
* chronic obstructive pulmonary disease who treated with inhaled β2 agonist
* significant kidney disease with eGFR <30%
* severe uncontrolled electrolyte abnormalities
* prior allergic reaction to Salbutamol
* Pregnancy and nursing women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Changes in plasma level of N-terminal pro-BNP at twelve weeks relative to baseline pro-BNP. | 12 weeks from baseline pro-BNP assessment

SECONDARY OUTCOMES:
Adverse cardiovascular event: Death, ICD discharge, significant ventricular arrhythmias and hospitalization due to heart failure exacerbation | 12 weeks after baseline assessment
  Record events of death, ICD discharge and hospitalization due to heart failure exacerbation. Interrogate ICD memory for significant ventricular arrhythmias (ventricular tachycardia and ventricular fibrillation) that did not cause ICD discharge.
NYHA class changes | 12 weeks after baseline assessment
  We will assess NYHA functional class at baseline and after 12 weeks from the beginning of study medication.
Echocardiography parameters changes | 12 weeks after baseline assessment
  END-SYSTOLIC DIAMETER: _ _ _ MM END-DIASTOLIC DIAMETER: _ _ _ MM LVEF (SIMPSON'S) : _____% Left atrial diameter: ____MM Left atrial area:______cm2 dP/dT: ___32/∆t (mm Hg/msec) E/A: ___ E': ___ cm/s E/E': _____ E wave deceleration time:_____msec Isovolumic relaxation time (IVRT):_____msec
  Dimensionless myocardial performance index (MPI) (n<0.4) :
  MPI=(TST-ET)/ET TST- total systolic time -from the end of mitral inflow A wave to the beginning of mitral inflow E wave ET - ejection time - time from the beginning to the end of left ventricular outflow tract Doppler envelope
Minnesota Living with Heart Failure Questionnaire changes | 12 weeks after baseline assessment
  repeat Minnesota Living with Heart Failure Questionnaire assessment
Non-ventricular arrhythmias and electrolytes disturbances | baseline, 1 week, 4 weeks, 8 weeks and 12 weeks
  Plain ECG will be performed at the specified time intervals to detect asymptomatic non-ventricular arrhythmias (atrial fibrillation, atrial flutter, atrial premature beats, etc.) The venous blood will be drawn at the specified time intervals to follow closely after potassium levels (for timely detection of salbutamol induced hypokalemia and to correct accordingly), as well to monitor sodium levels as a prognostic and clinical marker of heart failure exacerbation

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin medical center, Petah Tikva, Israel